CLINICAL TRIAL: NCT01517529
Title: Evaluating the Role of the Immune Responses in the Emergence of HCV NS3 Resistance Mutations During Protease Inhibitor Therapy
Brief Title: Evaluating the Role of Immune Responses in the Emergence of Protease Inhibitor Mutations
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mohamed Tarek Shata, Principal investigator, University of Cincinnati
Other Study IDs: UC 11101915
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood lymphocytes from enrolled subjects will be retained until all investigations will be performed and publications are generated. After that remaining samples will be discarded properly according to the Biosafety instructions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 10 Hepatitis C infected subjects: 10 chronically HCV-infected patients who fail the standard peg-IFN and Ribavirin therapy (NR) and are therefore eligible for combined treatment with Protease Inhibitor therapy.

SUMMARY:
The major goal of this project is to identify the role of the immune responses in the emergence of protease inhibitor mutants during therapy.

DETAILED DESCRIPTION:
Objective 1: Evaluate the role of the immune responses in determining the emergence of HCV NS3 resistance mutation during protease inhibitor therapy

Hypothesis 1 (HT 1): Low HLA binding to peptides containing protease inhibitor resistance mutations is associated with the emergence of protease inhibitor mutants during therapy and failure of the treatment.

Hypothesis 2 (HT 2): A hole in T cell repertoire may allow emergence of protease inhibitor mutants during protease inhibitor therapy which leads to loss of the immune responses to these mutants and failure of treatment.

ELIGIBILITY:
Inclusion Criteria: All chronically HCV-infected patients who fail peg-IFN and RBV therapy and are eligible for combined treatment with PI therapy will be enrolled. Briefly, this includes:

1. Male or female
2. Age 18 to 65
3. Chronic HCV infection evidenced by liver biopsy or persistent HCV viremia for >6 months
4. Treatment experienced and classified as non-responder or relapser to prior interferon-based therapy.

Exclusion criteria:

1. Treatment naïve chronically HCV-infected patients.
2. Patients with a history of inflammatory bowel diseases (IBD) or suspected IBD, autoimmune diseases, including rheumatoid arthritis, and any patients on systemic immunomodulators.
3. Pregnancy
4. HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators plan to enroll 20 human subjects with chronic hepatitis C virus infection from the outpatient clinic at the University of Cincinnati College of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tarek. M Shata, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Abdel-Hameed EA, Rouster SD, Ji H, Ulm A, Hetta HF, Anwar N, Sherman KE, Shata MT. Evaluating the Role of Cellular Immune Responses in the Emergence of HCV NS3 Resistance Mutations During Protease Inhibitor Therapy. Viral Immunol. 2016 May;29(4):252-8. doi: 10.1089/vim.2015.0093. Epub 2016 Feb 17. PMID 26885675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We plan to enroll 10 chronically HCV-infected patients who fail the standard peg-IFN and Ribavirin (RBV) therapy (NR) and are therefore eligible for combined treatment with PI therapy according to the recent FDA approvals for Boceprevir. Patients will be recruited from the outpatient clinics at the University of Cincinnati College of Medicine
Groups:
- 10 Hepatitis C Infected Subjects: 10 chronically HCV-infected patients who failed the standard peg-IFN and Ribavirin therapy (NR) and are therefore eligible for combined treatment with Protease Inhibitor therapy.
Period: Overall Study
Arm/Group | 10 Hepatitis C Infected Subjects
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: chronically HCV-infected patients who fail the standard peg-IFN and Ribavirin (RBV) therapy (NR)
Arm/Group | 10 Hepatitis C Infected Subjects
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years]
  Responders | 55.3 (14.03)
  Non responders | 60.00 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Standard Treatment
Description: Blood samples will be drawn while the subject is on treatment to measure viral load and HCV-specific immune responses.
Time Frame: 9 months
Population: Measure HCV viral load and HCV-specific immune responses at baseline
Measure: Number; unit: participants
Arm/Group | 10 Hepatitis C Infected Subjects
Number analyzed (Participants) | 10
participants
  complete standard treatment | 10
  not complete | 0

2. Secondary Outcome: Number of Participants Who Cleared the Virus
Description: Blood samples will be drawn while the subject is on treatment to measure viral load and HCV-specific immune responses
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | 10 Hepatitis C Infected Subjects
Number analyzed (Participants) | 10
participants
  responder | 7
  Non-responder | 3

ADVERSE EVENTS:
Arm/Group | 10 Hepatitis C Infected Subjects
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Hepatitis C Infected Subjects (N=10)
Infection (Infections and infestations) | 1 (1) — Unrelated to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes